CLINICAL TRIAL: NCT04064840
Title: Gonadotrophin Releasing Hormone Agonist for Dual Trigger in in Vitro Fertilization and for Luteal Phase Support in Frozen-thawed Embryo Transfer
Brief Title: GnRH Agonist for Dual Trigger in IVF and for Luteal Phase Support in FET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 18-393; 06171626 (Other Grant/Funding Number: HMRF)
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Subfertility
Keywords: subfertility; IVF; FET; dual trigger; luteal phase support; Gonadotrophin releasing hormone agonist; live birth rate
MeSH Terms: conditions — Infertility | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IVF: dual trigger (Active Comparator): When at least three follicles reach 18 mm in diameter, recombinant hCG 0.25mg and decapeptyl 0.2mg will be injected subcutaneously.
  Interventions: Drug: IVF: Decapeptyl and hCG
- IVF: hCG trigger (Placebo Comparator): When at least three follicles reach 18 mm in diameter, recombinant hCG 0.25mg and normal saline will be injected subcutaneously.
  Interventions: Drug: IVF: hCG and normal saline
- FET: agonist (Active Comparator): On the day of FET, decapeptyl 0.1 mg will be injected subcutaneously.
  Interventions: Drug: FET: Decapeptyl
- FET: control (Placebo Comparator): On the day of FET, normal saline will be injected subcutaneously.
  Interventions: Drug: FET: Normal Saline

INTERVENTIONS:
Drug: IVF: Decapeptyl and hCG — When at least three follicles reach 18 mm in diameter, recombinant hCG 0.25mg and decapeptyl 0.2mg will be injected subcutaneously.
  Other Names: IVF: hCG
  Arms: IVF: dual trigger
Drug: FET: Decapeptyl — On the day of FET, decapeptyl 0.1 mg will be injected subcutaneously.
  Other Names: FET: normal saline
  Arms: FET: agonist
Drug: IVF: hCG and normal saline — When at least three follicles reach 18 mm in diameter, recombinant hCG 0.25mg and normal saline will be injected subcutaneously.
  Other Names: IVF: Decapeptyl and hCG
  Arms: IVF: hCG trigger
Drug: FET: Normal Saline — On the day of FET, normal saline will be injected subcutaneously.
  Other Names: FET: Decapeptyl
  Arms: FET: control

SUMMARY:
The objectives of this study are to compare the efficacy of the dual trigger group vs the hCG trigger group on the live birth rate in women undergoing IVF and the efficacy of the agonist in LP group vs the placebo group on the live birth rate in women undergoing FET.

DETAILED DESCRIPTION:
Trial design:

A randomised, double-blinded and placebo controlled trial will be performed in IVF cycles and another randomised, double-blinded and placebo controlled trial will be performed in FET cycles.

Treatment of subjects:

IVF Women being scheduled for IVF at Department of Obstetrics & Gynaecology of Kwong Wah Hospital and Queen Mary Hospital will be assessed for eligibility. Eligible women will be recruited for the study and each woman will only be included in the study. Informed written consent will be obtained after counseling.

All techniques of IVF including ovarian stimulation, harvesting of oocytes, insemination with specially prepared sperm and embryo culture in the laboratory will be according to local protocols. Women will receive ovarian stimulation using antagonist protocol. Ultrasound scanning will be arranged on day 2-3 of menses for the antral follicle counts and to exclude the presence of ovarian cyst. Oestradiol and progesterone concentration will be checked and if they are basal, ovarian stimulation with gonadotropin injections will be given. GnRH antagonist will be started on day 6 of ovarian stimulation. Regular ultrasound monitoring will be performed to monitor the growth of follicles. Adjustment of the gonadotropin dosage is corresponding to the number and size of follicles.

Randomization When three follicles reach 18 mm in diameter, recruited women will be randomized according to a computer-generated randomization list prepared by a designated research nurse into one of the following: (1) the dual trigger: recombinant hCG 0.25mg and decapeptyl 0.2mg subcutaneously and (2) the hCG trigger: recombinant hCG 0.25mg subcutaneously and normal saline.

Transvaginal ultrasound-guided egg retrieval will be scheduled 36 hours after the dual or hCG trigger. Intracytoplasmic sperm injection will be performed if necessary, depending on the semen quality of the husbands. A maximum of 2 embryos or blastocysts will be replaced 2 days or 5 days after egg retrieval according to the standard protocol under transabdominal ultrasound guidance.

Two days after egg retrieval, each woman will receive vaginal progesterone (Endometrin 100mg bd) for two weeks for the luteal phase support.

FET Women being scheduled for FET will be assessed for eligibility. Eligible women will be recruited for the study and each woman will only be included in the study with one FET cycle. Informed written consent will be obtained.

Women with regular ovulatory cycles will undergo the standard procedures of blood taking to identify the day of luteinizing hormone (LH) surge, which is defined as an elevation of the LH to 2 times the level of the average of the previous 3 days and the absolute level of the LH surge is greater than 20 IU/L. Transvaginal ultrasound will be done to measure the endometrial thickness on the day after the LH surge. A maximum of two early cleavage embryos or two blastocysts will be transferred 3 days or 6 days after the LH surge respectively.

Randomization On the day of FET, recruited women will be randomized into one of the following two groups: (1) decapeptyl 0.1 mg subcutaneously and (2) normal saline as control group according to a computer-generated randomization list prepared by a designated research nurse.

The rest of the embryo transfer procedure will be the same as our usual practice.

Blinding The women and the physicians will not know the group allocation. Only the research nurse will know the group allocation, but they will not be involved in the patient care.

Follow-up and data collection A urine pregnancy test is performed 18 days after the dual or hCG trigger in IVF cycles or the LH surge in FET cycles. If the pregnancy test is positive, transvaginal ultrasound will be performed 2 weeks later to locate the pregnancy and foetal viability. Subsequent management will be the same as other women with early pregnancy. They will be referred for antenatal care when the pregnancy is on-going at 8-10 weeks.

Follow-up Written consent regarding retrieval of pregnancy and delivery data from both public and private sectors will be sought from the patient at the time of study. The obstetric outcomes will be traced from the electric patient record system if the patients deliver in Hospital Authority hospitals. A pre-formatted letter with replying address available will be given to the patient at the end of the study period and is to be filled by the private obstetrician and returned to us after delivery. If no reply letter is received 2-3 months after the expected date of confinement of the patient, a letter including patient's authorization will be sent to the corresponding private obstetrician to retrieve the information of the pregnancy outcomes. The outcome of the pregnancy (delivery, miscarriage), number of babies born, birth weights and obstetrics complications will be recorded.

ELIGIBILITY:
IVF

Inclusion criteria:

- Women aged <43 years at the time of IVF treatment

Exclusion criteria:

* Preimplantation genetic diagnosis treatment
* Use of donor oocytes or donor embryos
* Hydrosalpinx shown on pelvic scanning and not surgically treated
* Women at risk of OHSS

FET

Inclusion criteria:

* Women aged <43 years at the time of IVF treatment
* Replacing early cleavage embryos or blastocysts after thawing
* FET in natural cycles

Exclusion criteria:

* Frozen early cleavage embryos thawed and cultured to blastocysts prior to transfer as requested by the patient
* Preimplantation genetic diagnosis treatment
* Use of donor oocytes or donor embryos
* Hydrosalpinx shown on pelvic scanning and not surgically treated

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 784 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | after 22 weeks
  delivery after 22 weeks

SECONDARY OUTCOMES:
Pregnancy | 18 days after the dual or hCG trigger in IVF cycles or the LH surge in FET cycles
  positive urine pregnancy test
Clinical pregnancy | 6 weeks
  presence of intrauterine gestational sac on ultrasound
Biochemical pregnancy | before 6 weeks
  positive urine pregnancy test not followed by clinical pregnancy
Ongoing pregnancy | 8 weeks
  viable pregnancy beyond gestation 8 weeks
Implantation rate | 1 day
  number of gestational sacs per embryo transferred
Adverse events | 8 weeks
  Ovarian hyperstimulation syndrome
Neonatal outcome | 40 weeks
  Birth weight of babies

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China